CLINICAL TRIAL: NCT00242892
Title: Prospective Study Randomized Multicentric On the Optimization Of the Installation Of Stent By Measurement Of the Intra-Coronary Pressure
Brief Title: FROST 4: Study of the Optimal Spreading of a Coronary Stent Guided With Pressure Into the Coronary Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Volcano Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P001003
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2007-03

CONDITIONS: Coronary Artery Insufficiency
Keywords: Deployment stent optimisation; Fractional Flow Reserve; Stent; Restenosis; Coronary

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Intra coronary measures of pressure
  Interventions: Procedure: Intra coronary measures of pressure

INTERVENTIONS:
Procedure: Intra coronary measures of pressure — Intra coronary measures of pressure

SUMMARY:
Hypothesis : it is known that the stent must be well opened out in order to avoid restenosis into the stent. Intra coronary pressure would allow the stent to be well deployed and so the restenose into the stent should diminish.

Primary purpose : this study intend to test the hypothesis of optimal spreading of coronary stent guided with pressure into coronary arteritis comparing 2 strategies with patients having a coronary procedure with stent, excluded patients with myocardial infarction.

DETAILED DESCRIPTION:
It is a randomized study, intending to treat, comparing the optimisation of the opening out of a stent into a coronar artery either guided with angiographic images only or with the assistance of pressure measurements plus angiographic control.

Several French centers participate to demonstrate superiority of one strategy. The criterion of principal judgement is the whole of cardiac events, criterion made up with the cardiac death, myocardial infarction, revascularisation by coronary bridging and/or angioplasty and positivity of the effort test.

Secondary criterions are :

* comparing cost to efficacy of the two strategies
* evaluating the angiographic restenosis into an under group of 200 patients (100 patients into each group)
* determining the optimal threshold of measurement of intra coronary pressure in a multicentric population
* comparing the ability of the different stents used to optimised the intra coronary pressure measurements

ELIGIBILITY:
Inclusion Criteria:

* patient sent to coronal angioplasty with putting of an active stent to treat a restenosis

Exclusion Criteria:

* acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2001-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The first group of patients will have a coronary procedure with stent and his good deployment will be controlled with angiographic images | during de study
  The first group of patients will have a coronary procedure with stent and his

SECONDARY OUTCOMES:
At 6 months cardiac events will be registered: patients will undergo a scintigraphic and effort test with thallium and a clinical exam | during the study
  At 6 months cardiac events will be registered: patients will undergo a
At 12 and 18 months they will undergo a clinical exam and cardiac events will be registered | during the study
  At 12 and 18 months they will undergo a clinical exam and cardiac events will be registered
Complementary examination | during the study
  Complementary examination

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LAFONT, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- European Georges Pompidou's Hospital, Paris, France